CLINICAL TRIAL: NCT06894420
Title: Comparison of Postoperative Analgesic Efficacy of Ultrasonographic Bilateral TAP (Transversus Abdominis Plane) Block and Anesthetic Infiltration Into Preperitoneal and the Surgical Field in Laparoscopic Unilateral TEP (Total Extraperitoneal) Herniorraphy
Brief Title: Comparison the Analgesic Efficacy of Ultrasonographic Bilateral TAP and Anesthetic Infiltration Into the Surgery Field for Laparoscopic Unilateral TEP Herniorrhaphy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine OZCAN, Assistant Investigator, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AC2122
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Laparoscopic Surgery; Herniorrhaphy; Inguinal Hernia Unilateral; Transversus Abdominis Plane (TAP) Block; Postoperative Analgesia
Keywords: Laparoscopic surgery; Inguinal hernia; postoperative analgesia; Transversus Abdominis Plane (TAP) Block
MeSH Terms: conditions — Bites and Stings; Hernia, Inguinal | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Prospective Randomize
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery Block (Active Comparator): After obtaining informed consent from the volunteer patients before surgery, the patients will be taken to the operating room, monitored and put to sleep with the general anesthesia procedure that we routinely apply in laparoscopic surgeries. In laparoscopic hernia repairs, patients will be placed in supine position, after appropriate aseptic conditions are provided (the surgical area will be wiped with 10% povidone iodine so that there is no dry area and covered with sterile green drapes). Under general anesthesia, a 1 cm incision will be made 1 cm inferior to the umbilical border, a 10 mm trocar will be inserted into the preperitoneal space and blunt dissection will be performed with a 30 degree camera. After observing the preperitoneal space, two 5 mm working trocars will be placed in the midline 2 cm and 6 cm inferior to the symphysis pubis. The cord structures and Cooper ligament will be exposed and the hernia sac will be freed from the anatomical structures of the cord. Prolene
  Interventions: Procedure: Surgeon-Initiated Local Anesthetic
- TAP Block (Active Comparator): Group-II patients will undergo bilateral TAP block under ultrasound guidance by the anesthesiologist before the patient wakes up after the operation is completed and the skin is sutured. During the block, a Hitachi brand linear USG probe will be sterilized and placed between the iliac wing and costae parallel to the costal margin in the mid-axillary line. Anatomically, skin, subcutaneous tissue, external oblique muscle, internal oblique muscle and transversus abdominis muscle will be visualized. Under USG guidance, a 21G 80 or 100 mm block needle will be advanced from medial to lateral (or lateral to medial) to reach the fascial plane between the internal oblique and transversus abdominis muscles. After confirming the block site by injecting 1-2 ml of 0.09% NaCl after negative aspiration, 15-20 ml (40-50 mg in each quadrant of the abdomen since the block will be performed bilaterally) of bupivacaine 0.5% concentration will be given to the patients in a controlled manner by negative as
  Interventions: Procedure: Transversus abdominis plane (TAP) block

INTERVENTIONS:
Procedure: Surgeon-Initiated Local Anesthetic — In laparoscopic hernia repairs, patients are positioned supine, and the surgical area is cleansed with povidone iodine and covered with sterile green drapes. A 1-centimeter incision will be made 1 centimeter below the umbilical border. A 10-mm trocar will be inserted into the preperitoneal space. The operation was filmed from the front with a 30-degree camera. After observing the preperitoneal space, two five-mm working trocars will be placed midline, two and six centimeters inferior to the symphysis pubis. Next, the cord structures and Cooper ligament will be exposed and the hernia sac freed from surrounding anatomical structures.Prolene mesh will be spread over the preperitoneal area to cover all hernia defects and secured to the Cooper ligament and abdominal wall with an absorbable fixation device. Group 1 patients undergo desufflation via 50 mg of bupivacaine into the preperitoneal space, followed by 10 mg of bupivacaine into each trocar incision and skin closure with sutures.
  Arms: Surgery Block
Procedure: Transversus abdominis plane (TAP) block — After the surgery, the anesthesiologist will use a TAP block under ultrasound guidance. Before the patient wakes up, the Hitachi ultrasound probe will be sterilized and positioned between the iliac wing and the costae. An ultrasound shows the skin, fat beneath it, the six abdominal muscle layers, and a support muscle.A thin needle goes through the skin from one side to the other to reach the muscle layers. The location of the block is confirmed by injecting 1-2 ml of 0.09% NaCl followed by negative aspiration. Patients receive 15-20 ml (40-50 mg per quadrant) of bupivacaine 0.5% concentration in a controlled manner with negative aspiration every 5 ml. The block is performed bilaterally.
  Arms: TAP Block

SUMMARY:
Laparoscopic inguinal hernia repair is a common surgical procedure, but postoperative pain management remains a challenge. This prospective, randomized study aims to compare the analgesic efficacy of preperitoneal and surgical site anesthetic infiltration with ultrasound-guided bilateral transversus abdominis plane (TAP) block in patients undergoing laparoscopic unilateral total extraperitoneal (TEP) herniorrhaphy. Sixty patients will be randomly allocated into two groups: Group-I will receive preperitoneal and surgical site infiltration with bupivacaine, while Group-II will receive ultrasound-guided bilateral TAP block with bupivacaine. The primary outcomes will be postoperative pain scores assessed using the visual analog scale (VAS) and additional analgesic requirements. Secondary outcomes will include postoperative hospital stay duration and cost-effectiveness. Demographic data, ASA scores, comorbidities, and operation times will be recorded. Postoperative pain will be managed with a multimodal approach, including paracetamol and NSAIDs. Rescue analgesia will be provided with intravenous paracetamol. Statistical analysis will be performed using t-tests, ANOVA, Wilcoxon-Mann-Whitney tests, and chi-square tests, as appropriate. This study aims to determine the optimal and most beneficial method for postoperative pain management and patient comfort following laparoscopic inguinal hernia repair.

DETAILED DESCRIPTION:
Abdominal fascial plane blocks are now considered adequate and reliable methods for the management of postoperative pain following both open and laparoscopic abdominal procedures. Abdominal fascial plane blocks have become an indispensable part of postoperative multimodal analgesia due to their cost-effectiveness, ease of use and relatively low complication rates since the introduction of ultrasound guidance. Although the type of pain after laparoscopy is different from laparotomy, mostly parietal pain (abdominal wall origin), patients also complain of visceral pain due to pneumoperitoneum. Many analgesic procedures are used as part of multimodal analgesia for postoperative pain, including nonsteroidal anti-inflammatory drugs (NSAIDs), opioids and regional anesthesia procedures. Regional anesthesia techniques in abdominal surgery include epidural analgesia, paravertebral block and transversus abdominis plan (TAP) block, quadratus lumborum block, transversalis fascial plan block, rectus sheath block. Inguinal hernia repair is one of the most common operations performed in general surgery clinics. Regardless of the etiology and type, surgical repair is considered the definitive treatment for inguinal hernia. The need for analgesic medication after laparoscopic repair of inguinal hernia is greatly reduced because the procedure reduces postoperative pain. The preperitoneal space and trocar incisions are two potential sites of pain in the laparoscopic total extraperitoneal (TEP) procedure. The TAP block, one of the truncal blocks, has been used in many studies in the literature for pain palliation after abdominal surgery.The transversus abdominis plane (TAP) block is a regional anesthetic technique that provides effective analgesia to the skin and muscles of the anterior abdominal wall as well as the parietal peritoneum. The TAP block is applied in the fascial plane between the internal oblique and transversus abdominis muscles. It targets the T6-L1 somatic nerves traveling in this plane. Currently, various techniques are used to perform TAP blocks, including the blind double POP technique, ultrasound-guided and laparoscopic-assisted approaches. Preperitoneal and surgical site local anesthesia can be performed effectively for postoperative analgesia in laparoscopic surgeries with laparoscopic visualization by the surgical team. Opioids are also the most commonly used narcotic analgesics for postoperative pain. Patients often require opioids for pain relief in the perioperative period, especially in abdominal surgery. However, the use of opioids can lead to a variety of side effects including excessive sedation, postoperative nausea, vomiting, urinary retention, constipation, hyperalgesia, respiratory depression and immunosuppression. Opioids may have various effects on immune function, such as modulation of cytokines, interaction with immune cells, affecting the neuroendocrine system and vascular permeability, and may contribute to postoperative complications such as infections and delayed wound healing due to increased inflammatory response. May prolong hospitalization. In order to reduce postoperative opioid consumption and opioid-related side effects, ultrasound-guided trunk block techniques have been developed and are now widely used in abdominal surgeries. Ultrasound-guided transversus abdominis plan block (TAPB) is an effective analgesic method used in anesthesia together with multimodal analgesia techniques.

In this study, we planned to compare the effects of laparoscopic preperitoneal and surgical site anesthetic infiltration and ultrasound-guided bilateral TAP block in laparoscopic herniorrhaphies in terms of postoperative pain scores and need for additional analgesics as the primary objective and postoperative hospital stay and cost as secondary objectives.In this study, patients will be asked preoperatively whether they would like to have a block for postoperative pain. Then they will be classified according to the block randomization method. Patients will be divided into 2 groups and will be named as Group-I and Group-II. After obtaining informed consent from the volunteer patients before surgery, the patients will be taken to the operating room, monitored and put to sleep with the general anesthesia procedure that we routinely apply in laparoscopic surgeries. In laparoscopic hernia repairs, patients will be placed in supine position, after appropriate aseptic conditions are provided (the surgical area will be wiped with 10% povidone iodine so that there is no dry area and covered with sterile green drapes). Under general anesthesia, a 1 cm incision will be made 1 cm inferior to the umbilical border, a 10 mm trocar will be inserted into the preperitoneal space and blunt dissection will be performed with a 30 degree camera. After observing the preperitoneal space, two 5 mm working trocars will be placed in the midline 2 cm and 6 cm inferior to the symphysis pubis. The cord structures and Cooper ligament will be exposed and the hernia sac will be freed from the anatomical structures of the cord. Prolene mesh will be spread over the preperitoneal area to cover all hernia defects and Prolene mesh will be fixed to the Cooper ligament and abdominal wall with absorbable fixation device. At this stage, in Group-I patients, the surgical field will be desuflated by injecting 50 mg bupivacaine into the preperitoneal space. Then, 10 mg bupivacaine will be injected into each trocar incision and the skin will be closed with sutures. Group-II patients will undergo bilateral TAP block under ultrasound guidance by an anesthesiologist before the patient wakes up after the operation is completed and the skin is sutured. During the block, Hitachi brand linear USG probe will be sterilized and placed between the iliac wing and costae parallel to the costal margin in the mid-axillary line. Anatomically, skin, subcutaneous tissue, external oblique muscle, internal oblique muscle and transversus abdominis muscle will be visualized. Under USG guidance, a 21G 80 or 100 mm block needle will be advanced from medial to lateral (or lateral to medial) to reach the fascial plane between the internal oblique and transversus abdominis muscles. After confirming the block site by injecting 1-2 ml of 0.09% NaCl after negative aspiration, 15-20 ml (40-50 mg in each quadrant of the abdomen since the block will be performed bilaterally) of bupivacaine 0.5% concentration will be given to the patients in a controlled manner by negative aspiration at every 5 ml. At the end of the operation, Parol 1 g i.v. and NSAID (Tenoxicam 20 mg i.v.) will be administered to the patients within the scope of multimodal analgesia without waking them up at the end of the operation, and the patients will be checked with VAS (visual analog scale) score within the first 24 hours after waking up and postoperative pain and analgesic need (if needed as postoperative analgesic, only Parol 1 gr. I.v.) will be evaluated. The aim of our study is to show the postoperative analgesic efficacy of preperitoneal and surgical site local anesthetic infiltration and USG-guided bilateral TAP block in patients undergoing laparoscopic hernia repair and whether they are superior to each other on postoperative pain. To find the most optimal and beneficial one in terms of patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients,
* She will undergo laparoscopic hernia repair surgery,
* ASA-I-II,
* Between the ages of 18 and 65,
* No history of anticoagulant or antiaggregant drug use,
* Regional anesthesia is not contraindicated and the anesthesiologist deems -appropriate for regional anesthesia,
* Under general anesthesia and will undergo laparoscopic surgery,
* Fully oriented and cooperative,
* Unilateral inguinal hernia,
* No previous surgery for inguinal hernia,
* No incision in the lower abdomen,
* Not using alcohol and drugs,
* No preoperative pain and
* Patients without symptoms of strangulated hernia will be included in the study.

Exclusion Criteria:

* Patients without consent
* Regional anesthesia is contraindicated,
* Those who will undergo open abdominal surgery,
* Not in the appropriate age range,
* Chronic diseases such as uncontrolled DM and HT,
* Drug allergy,
* Taking anticoagulant or antiaggregant drugs,
* History of chronic analgesic use,
* Presence of active infection in the area to be blocked,
* Will not be able to comply with postoperative pain /VAS follow-up,
* Patients with ASA-III-IV,
* Patients with bilateral inguinal and scrotal hernias,
* Patients who have been previously operated for inguinal hernia and have an incision in the lower abdomen,
* Those with a history of alcohol and drug abuse
* Preoperative pain and
* Those with symptoms of strangulated hernia will not be included in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 24 hours
  Visual Analog Scale. It will be used to assess postoperative pain. The degree of pain of the patient will be evaluated with a scoring scale from 1 to 10. 0- No pain...... 10- Intolerable pain.

CONTACTS AND LOCATIONS:
Overall Officials: EMINE OZCAN, MD, Study Director — Başakşehir Çam ve Sakura Şehir Hastanesi
Locations (1):
- Başakşehir Çam ve Sakura Şehir Hastanesi, Başakşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 01.01.2026- 01.-1.2027
Access Criteria: The types of analyses that are appropriate for data sharing and the statistical methods for those analyses need to be approved by the independent reviewer.

REFERENCES:
- [Background] Mughal A, Khan A, Rehman J, Naseem H, Waldron R, Duggan M, Khan W, Barry K, Khan IZ. Laparoscopic-assisted transversus abdominis plane block as an effective analgesic in total extraperitoneal inguinal hernia repair: a double-blind, randomized controlled trial. Hernia. 2018 Oct;22(5):821-826. doi: 10.1007/s10029-018-1819-8. Epub 2018 Sep 1. PMID 30173291
- [Background] Colak S, Akkus O, Gurbulak B, Cakar E, Bektas H. Infiltration of bupivacaine into the preperitoneal space and trocar incisions of patients undergoing laparoscopic totally extraperitoneal repair of unilateral inguinal hernia: a prospective randomized controlled observational study. Wideochir Inne Tech Maloinwazyjne. 2020 Mar;15(1):11-17. doi: 10.5114/wiitm.2019.84385. Epub 2019 Apr 11. PMID 32117481
- [Background] Paasch C, Fiebelkorn J, De Santo G, Aljedani N, Ortiz P, Gauger U, Boettge K, Full SH, Anders S, Hunerbein M. Ultrasound-versus visual-guided transversus abdominis plane block prior to transabdominal preperitoneal ingunial hernia repair. A retrospective cohort study. Ann Med Surg (Lond). 2020 Sep 22;59:281-285. doi: 10.1016/j.amsu.2020.09.017. eCollection 2020 Nov. PMID 33133582
- [Background] Grape S, Kirkham KR, Albrecht E. The analgesic efficacy of transversus abdominis plane block vs. wound infiltration after inguinal and infra-umbilical hernia repairs: A systematic review and meta-analysis with trial sequential analysis. Eur J Anaesthesiol. 2022 Jul 1;39(7):611-618. doi: 10.1097/EJA.0000000000001668. Epub 2022 Feb 7. PMID 35131973
- [Background] Salmonsen CB, Lange KHW, Rothe C, Kleif J, Bertelsen CA. Cutaneous sensory block area of the laparoscopic-assisted transversus abdominis plane block. Dan Med J. 2024 Sep 9;71(10):A02240142. doi: 10.61409/A02240142. PMID 39323259
- See also: The National Center for Biotechnology Information advances science and health by providing access to biomedical and genomic information. — https://pubmed.ncbi.nlm.nih.gov/